CLINICAL TRIAL: NCT04962269
Title: Different Models of Multiple B-value DWI and Their Applications in Diagnosis of Prostate Cancer
Brief Title: Application of DWI in Diagnosis of Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2019176
Record Dates: First submitted 2021-06-29; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer; Benign Prostatic Hyperplasia
Keywords: benign prostatic hyperplasia; Diffusion weighted imaging
MeSH Terms: conditions — Prostatic Neoplasms; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- prostate cancer: The patient was pathologically diagnosed with prostate cancer
  Interventions: Diagnostic Test: MRI
- benign prostatic hyperplasia: The patient was pathologically diagnosed with benign prostatic hyperplasia

INTERVENTIONS:
Diagnostic Test: MRI — monoexponential model, intravoxel incoherent motion (IVIM) model and stretched exponential model
  Groups: prostate cancer

SUMMARY:
This study compared the performance of different models of multiple b-value DWI in diagnosing prostate cancer.

DETAILED DESCRIPTION:
Diffusion weighted imaging (DWI) plays an important role in the diagnosis and stratification of prostate cancer. Traditional DWI apply the apparent diffusion coefficient (ADC) to reflect the diffusion of tissue water, which is a parameter calculated by a monoexponential model with 2b values. In recent years, the development of multiple b-value DWI facilitates the appearance of many new mathematical models. Different models have different features, but their value of applications in prostate cancer still need to be confirmed. This study was aiming to: (1) compare the parameters derived from monoexponential model, intravoxel incoherent motion (IVIM) model and stretched exponential model between prostate cancer and benign prostatic hyperplasia; (2) compare the difference of these parameters between low-grade (Gleason score ≤ 3+4) and high-grade (Gleason score ≥ 4+3) cancer; (3) find whether these parameters derived from new models are superior to ADC derived from traditional monoexponetial model.

ELIGIBILITY:
Inclusion Criteria:

1. The exam including T1WI、T2WI and multiple b-value DWI.
2. Comfired by pathology as prostate cancer or benign prostatic hyperplasia in one month after the MRI exam.

Exclusion Criteria:

* 1.No Gleason score data. 2.Awful quality of imagings or artifacts affectting diagnosis. 3.No lesion larger than 0.5cm. 4.Any surgery or treatment before MRI exam. 5.Biopsy in 4 weeks before MRI exam.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with prostatic diseases confirmed as prostate cancer or benign prostatic hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2018-06-21 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
pathological diagnosis | 2013.10-2018.6
  prostate cancer or benign prostatic hyperplasia

CONTACTS AND LOCATIONS:
Overall Officials: Jianyu Liu, Study Director — Peking University

IPD SHARING:
Plan to Share IPD: No